CLINICAL TRIAL: NCT03038308
Title: Treatment of Hyperprolactinemia With the Non-ergoline Dopamine Agonist Ropinirole: A Dose Escalation Study of Efficacy and Tolerability
Brief Title: Treatment of Hyperprolactinemia With the Non-ergoline Dopamine Agonist Ropinirole
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAI8604; 1R21DK112093-01 (NIH)
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Hyperprolactinemia; Prolactinoma
Keywords: ropinirole; hyperprolactinemia; prolactin
MeSH Terms: conditions — Hyperprolactinemia; Prolactinoma | interventions — ropinirole

STUDY DESIGN:
Intervention Model Description: 1) Forced titration dose response PKPD study and 2) A prospective open-label outpatient dose escalation trial of ropinirole for treatment of prolactinomas and hyperprolactinemia.
Masking Description: Open-label studies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ROP Intervention (Experimental): Patients with hyperprolactinemia were treated with long-term ROP therapy for 6 months in an open-label dose escalation study
  Interventions: Drug: Ropinirole

INTERVENTIONS:
Drug: Ropinirole — 0.25mg/day - 6.0mg/day oral non-ergoline dopamine agonist ropinirole
  Other Names: ROP therapy

SUMMARY:
The purpose of this study is to evaluate the use of the non-ergoline dopamine agonist ropinirole for the treatment of hyperprolactinemia in patients with idiopathic hyperprolactinemia and prolactinomas.

DETAILED DESCRIPTION:
Treatment of prolactin secreting pituitary tumors with traditional ergot dopamine agonist drugs can be limited by medication side effects, pharmacologic resistance, and by concerns regarding the potential risk of cardiac valve disease. The overall goal of this project is therefore to evaluate, for the first time, the efficacy and tolerability of the selective D2/D3 receptor non-ergot dopamine agonist ropinirole for the treatment of prolactinomas. This proposal will establish the pharmacologic profile of this medication when used to treat hyperprolactinemia in patients with prolactinomas and will determine the impact of long-term ropinirole administration on critical clinical parameters including serum prolactin levels, gonadal function, and tumor regression, in order to establish ropinirole's utility as a new, clinically efficacious, safer and more tolerable therapeutic option for the treatment of prolactinomas that may prove particularly useful in patients with underlying cardiac valve disease and in those with resistance or intolerance to ergot dopamine agonists.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years
* Prolactin level (PRL) ≥2 times upper limit of normal
* Pituitary adenomas on MRI ≤ 1.5cm in greatest diameter and ≥ 5mm from the optic chiasm
* Normal renal and liver function
* Agrees to barrier contraception if pre-menopausal

Exclusion Criteria:

* Use of medications known to interfere with PRL secretion and PRL and Ropinirole (ROP) metabolism
* Use of another dopamine agonist during the 4 weeks prior
* Pituitary stalk compression on MRI
* History of visual field abnormalities or previous radiation
* Untreated hypothyroidism
* Consumption of > 2 alcoholic drinks per day
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Page-Wilson, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu S, Hu C, Peters J, Tsang A, Cremers S, Bies R, Page-Wilson G. Pharmacokinetics and pharmacodynamics of ropinirole in patients with prolactinomas. Br J Clin Pharmacol. 2019 Feb;85(2):366-376. doi: 10.1111/bcp.13802. Epub 2018 Nov 22. PMID 30362146

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 Subject was determined to be ineligible after consenting.
Period: Overall Study
Arm/Group | ROP Intervention
Started | 15
Completed | 11
Not Completed | 4
Not completed — Surgical resection | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Only 15 out of 16 enrolled subjects went on to receive study therapy; however, demographic information was collected for all 16 enrolled subjects.
Arm/Group | ROP Intervention
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Prolactin [Mean (Standard Deviation); unit: ng/mL] | 126 (41.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects That Achieved PRL Normalization as Defined by a Serum Prolactin Level Less Than 25ng/mL at Any Time Point During the Study Treatment Period.
Description: Serum prolactin concentrations (PRL levels) were measured in patients at baseline, 2 and 4 weeks after starting therapy and then once monthly thereafter for 24 weeks. Serum prolactin was measured in duplicate by two-site chemiluminescent enzyme immunometric assay using the Immulite 1000 Analyzer (Siemens Healthcare Diagnostics, Deerfield, IL). The reference range for serum prolactin is 1.9-25 ng/ml for adult females.
Time Frame: 6-12 months
Population: Of the 16 subjects enrolled, 1 was deemed ineligible after completion of screening, 2 relocated out of state prior to taking first dose, 1 was withdrawn after week 1 following decision to pursue surgical resection of the prolactinoma. 12 participated longitudinally -- 1 was lost to follow-up after 16 weeks; 11 subjects completed 24 weeks and 5/11 subjects continued ropinirole therapy for one year with 2/11 remaining in protocol for 17 months due pandemic related delays in final visits.
Measure: Count of Participants; unit: Participants
Arm/Group | ROP Intervention
Number analyzed (Participants) | 12
Participants | 6

2. Secondary Outcome: Number of Subjects With Stable or Decreased Tumor Size
Description: Number of subjects with stable or decreased tumor size from baseline assessment to assessment after 6 months of treatment. Radiologic assessment of tumor size before and after treatment will be made by MRI.
Time Frame: 6 months
Population: Nine participants analyzed as only 9 participants had a followup MRI at 6 months.
Measure: Number; unit: participants
Arm/Group | ROP Intervention
Number analyzed (Participants) | 9
participants | 7

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ROP Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ROP Intervention (N=10)
Fatigue (General disorders) | 6
Nausea (General disorders) | 4
Headache (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03038308/Prot_SAP_000.pdf